CLINICAL TRIAL: NCT00679692
Title: Insulin-Like Growth Factor-1,Insulin-Like Growth Factor Binding Protein-3 and Human Growth Hormone in Serum of Patients With Chronic Liver Disease and Possible Clinical Applications.
Brief Title: Evaluation the Growth Factors(IGF-1,IGFBP-3and HGH)in Patients With Chronic Liver Disease
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Kaoshing Medical University Chung-Ho Memorial Hospital, Kaoshing Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUH-IRB-950123; KMUH-IRB-950123
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2006-01

CONDITIONS: Hepatitis; Liver Cirrhosis; Hepatocellular Carcinoma
Keywords: GH,IGF-1, IGFBP-3
MeSH Terms: conditions — Hepatitis; Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 3:: three arms for study

SUMMARY:
BACKGROUND The insulin-like growth factor system (IGFs) plays an important role in cell growth and differentiation. Nevertheless, the roles played by insulin-like growth factor-1 (IGF-1), insulin-like growth factor binding protein-3 (IGFBP-3) and human growth hormone (HGH) in the progression of chronic liver disease remain to be elucidated and investigated.

METHODS The subjects in the present study included 60 healthy controls, 30 hepatitis patients, 60 liver cirrhosis patients and 60 untreated hepatocellular carcinoma patients. Blood was drawn by venipuncture into Venoject tubes. To find the possible correlations between liver damage and IGFs, serum IGF-1, GH, IGFBP-3 concentration and related biochemical parameters were measured. We used immunoradiometric assay to determine the levels of IGF-1, HGH and IGFBP-3 in serum.

DETAILED DESCRIPTION:
healthy controls:one blood sample (7.5 cc) hepatitis: three blood samples, at admission, at 3rd and 7-10th day of admission liver cirrhosis: two blood samples, at 1-2 years interval (7.5 cc/each session) hepatocellular carcinoma: three blood samples, before, 1 day after and at the 7th day of transcatheter arterial chembolizatiom

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hepatocellular carcinoma
* Must be primary Hepatocellular carcinoma and untreament

Exclusion Criteria:

* treatment Hepatocellular carcinoma

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute hepatitis liver cirrhosis hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: chiou m Lin, Ms, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Division of Radio immunoassay lab,Department of Nuclear Medical University Hospital,No.100 Tzyou 1st Road, Kaohsiung City, Taiwan